CLINICAL TRIAL: NCT01635270
Title: Randomized Phase 2 Study Evaluating the Interest of Mid-position Strategy Versus ITV (Internal Target Volume) Strategy in Radiotherapy Treatment for Patients With a Locally Advanced Non-resected Non-small Cell Lung Carcinoma (NSCLC).
Brief Title: Phase 2 Study Evaluating Mid-position Strategy in Radiotherapy Treatment for Patients With a Locally Advanced Non-small Cell Lung Carcinoma
Acronym: midP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: CREATIS Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: midP; 2012-A00413-40 (Other: ANSM number); ET12-033 (Other: Sponsor ID)
Record Dates: First submitted 2012-06-29; First posted 2012-07-09 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer; Radiation Therapy; Locally Advanced Disease; Non-metastatic Disease; Non-resectable Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midP arm (Experimental): Patients treated with midP radiotherapy strategy.
  Interventions: Radiation: mid-position radiation strategy
- ITV arm (Active Comparator): Patient treated with radiotherapy ITV strategy
  Interventions: Radiation: ITV

INTERVENTIONS:
Radiation: mid-position radiation strategy — The midP strategy defines the target as the time weighted average tumor position (mid-position) plus an additional margin, computed specifically for each patient, that takes into account the tumor motion in each direction. This strategy can help to safely reduce toxicity while preserving treatment efficacy
  Arms: midP arm
Radiation: ITV — The ITV strategy is the conventional one. It consists in defining the target as the volume covering the whole tumor motion.
  Arms: ITV arm

SUMMARY:
The purpose of this study is to establish on the market and to clinically evaluate a new strategy of treatment for patients with locally advanced non-small cell lung cancer using deformable repositioning of 4D imaging.

ELIGIBILITY:
Inclusion Criteria:

* patient with a NSCLC, non-resected, non-metastatic including a parenchyma portion
* Age >= 18 years
* PS <=2
* CT-scan within 3 months at inclusion
* PET-scan within 3 months at inclusion
* Respiratory functional exploration within 3 months at inclusion
* estimated V20 (by radiotherapist)< 35% on conventional pre-radiotherapy imaging
* Tumor T0 to T4, M0; N1, N2 ou N3 by isolateral supra-clavicular involvement
* Measurable disease according to RECIST criteria 1.1
* Curative intent Chest conventional radiation therapy
* Radiation indication validated by a multidisciplinary meeting
* Adequate contraceptive method for the whole study duration and for up to 28 days after the end of radiation
* Mandatory affiliation with a health insurance company
* Patients must provide dated & written consent

Exclusion Criteria:

* Prior surgery for NSCLC
* NSCLC nearby pulmonary apex or strictly intra-thoracic with no intra-parenchyma portion
* Metastatic disease or N3 contralateral lymph node
* History of chest irradiation
* History of known increased intrinsic radiosensibility
* Hypersensibility to active substance or excipient of fluoro-deoxyglucose-18F
* Life expectancy < 6 months
* Patient with a concurrent malignancy or with a history of malignancy (excepted adequately treated basal cell skin carcinoma or cervical squamous cell carcinoma or other malignancies free of the disease for at least 5 years)
* Pregnant or breastfeeding women
* Psychological, sociological or geographical conditions that would limit compliance with study requirements
* Patient deprived of freedom
* Patient has concomitant participation to an other investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
1 year Progression Free Survival rate | 1 year
  Efficacy evaluation of the midP strategy in comparison with ITV strategy in patient with locally advanced, non-resected NSCL cancer treated with radiotherapy

SECONDARY OUTCOMES:
Local tumor control rate | 1 year and 2 years after the end of irradiation
Overall survival | 1 year and 2 years post irradiation
To determine acute and late pulmonary toxicity in the 2 arms, including respiratory functional exploration | Week1; Week 2; Week3; Week4; Week5; Week6; Week7 during the radiation, then 4 weeks, 3 months; 6 months ,one year and 2 years after the irradiation beginning

CONTACTS AND LOCATIONS:
Overall Officials: Line CLAUDE, MD, Principal Investigator — Centre Léon Bérard, Lyon, FRANCE
Locations (1):
- Centre Léon Bérard, Lyon, France